CLINICAL TRIAL: NCT00596557
Title: Phase IV: Effect of Everolimus and CNI Minimalization on Renal Function.
Brief Title: Everolimus and Low Dose CNI Compared With MMF and Full CNI Dose in Heart Transplanted Patients: One Year Follow up
Acronym: CRAD001AILO2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Tuvia Ben Gal MD, Director of the heart failure unit, Cardiology department, Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 004765
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Rejection of Cardiac Transplant
Keywords: Renal function, heart transplant, everolimus
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus, Immunosupression (Experimental): everolimus and reduced dose CNI: reduced dose CNI (cyclosporine level of 50-100)with everolimus levels of 3-8.
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — reduced dose CNI (cyclosporine level of 50-100)with everolimus levels of 3-8.
  Other Names: certican

SUMMARY:
The different mechanisms of action of Everolimus and cyclosporine suppress immune function in synergistic manner. Thus it is postulated that the use of Everolimus in combination with cyclosporine permits a significant cyclosporine dose reduction without loss of immunosuppressive activity in the clinical setting.

The aim of the present study is to evaluate the evolution of renal function after initiation of Everolimus and minimalisation of CNI dose.

DETAILED DESCRIPTION:
Everolimus is a new proliferation signal inhibitor with immunosuppressive and antiproliferative activity.

The mechanism of action of Everolimus is distinct from that of calcineurin inhibitors.

Cardiac allograft vasculopathy is the major cause of late death in cardiac transplant patients.

The different mechanisms of action of Everolimus and cyclosporine suppress immune function in synergistic manner. Thus it is postulated that the use of Everolimus in combination with cyclosporine permits a significant cyclosporine dose reduction without loss of immunosuppressive activity in the clinical setting.

The aim of the present study is to evaluate the evolution of renal function after initiation of Everolimus and minimalisation of CNI dose.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Signed informed consent
* 6 months to 15 year after heart transplantation
* Stable heart allograft function without rejection for at least 12 months
* Same immunusuppressive drugs for at least 3 months
* CNI based immunusuppression, with Cyclosporin levels C0 100-200 ng/ml FK levels of 5-10 ng/ml for preserved CNI levels.
* Poor renal function: creatinine > 1.5 mg%.

Exclusion Criteria:

* Suspected non-compliance
* Intolerance to Everolimus
* Life expectancy < 1year
* Proteinuria > 1.5 g/24u/1.73m2
* Previous sirolimus treatment
* Patients who received any other investigational drug
* Patients with platelet count <50,000/mm³ before baseline.
* Presence of severe hypercholesterolemia (≥350 mg/dL; ≥9 mmol/L) or hypertriglyceridemia (≥750 mg/dL; ≥8.5 mmol/L)
* Patients with an absolute neutrophil count of ≤ 1,500/mm3 or white blood cell count of ≤ 4000/mm³ at baseline
* Patients with a known hypersensitivity to similar drugs and to the components of the formulations
* Patients being treated with terfenadine, astemizole, or cisapride.
* Patients who are treated with drugs strong inducers or inhibitors of cytochrome P450 3A4.
* Patients with any past (within the past 5 years) or present malignancy (other than excised basal cell carcinoma)
* Patients with clinically significant systemic infection.
* Existence of any surgical or medical condition, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and excretion of study medication, and/or the presence of severe diarrhea or active peptic ulcer.
* Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evolution of renal function after initiation of Everolimus and minimalisation of CNI dose. | 1 year

SECONDARY OUTCOMES:
The occurrence of major adverse cardiovascular events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tuvia Ben Gal, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Cardiology Department, Rabin Medical Center, Petah Tikva, Petah Tikva, Israel